CLINICAL TRIAL: NCT00109863
Title: Phase II Trial of Hu14.18-IL2 (EMD 273063) in Subjects With Advanced Melanoma
Brief Title: Hu14.18-Interleukin-2 Fusion Protein in Treating Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000426431; P30CA014520 (NIH); CO04601 (Other: University of Wisconsin Carbone Cancer Center); NCI-6304; H-2004-0396 (Other: Institutional Review Board); NCI-2009-00051 (Registry Identifier: NCI Trial ID); A533300 (Other: UW Madison); R01CA032685 (NIH); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2015-02

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — lorukafusp alfa

ARMS (1):
- Hu14.18-IL2 Treatment (Experimental): Hu14.18-IL2 will be given on days 1, 2, and 3 of each course of therapy as a 4 hour continuous IV infusion at a daily dose of 6 mg/m2. Treatment courses will be repeated every 28 days at the same dose.
  Interventions: Biological: hu14.18-IL2 fusion protein

INTERVENTIONS:
Biological: hu14.18-IL2 fusion protein

SUMMARY:
RATIONALE: Biological therapies, such as hu14.18-interleukin-2 fusion protein, may stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase II trial is studying how well hu14.18-interleukin-2 fusion protein works in treating patients with advanced melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical antitumor activity of hu14.18-interleukin-2 fusion protein in patients with advanced melanoma.
* Determine the duration of response in patients treated with this drug.

Secondary

* Determine the adverse events in patients treated with this drug.
* Determine the in vivo immunologic activation in patients treated with this drug.
* Determine the induction of anti-hu14.18 and anti-interleukin-2 antibodies in patients treated with this drug.
* Determine tumor antigen recognition by this drug in select patients with cutaneous metastatic tumors, as measured by binding of the drug to the cutaneous metastatic tumor and microscopic changes (including immune cell density and phenotype) of the tumor tissue.

OUTLINE: Patients receive hu14.18-interleukin-2 fusion protein IV over 4 hours on days 1-3. Treatment repeats every 28 days for 2 courses in the absence of symptomatic disease progression or unacceptable toxicity. Patients then undergo disease reassessment. Patients with an objective partial or complete clinical response or stable disease receive 2 additional courses of treatment.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 7-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Advanced disease
* Measurable disease by clinical assessment or imaging
* No known standard curative therapy exists

  * Disease no longer controlled by surgery, chemotherapy, or radiotherapy
* No clinically detectable pleural effusion or ascites
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,500/mm^3 OR
* Granulocyte count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL

Hepatic

* AST and ALT < 2 times normal
* Bilirubin < 2.0 mg/dL
* Hepatitis B surface antigen negative
* No clinical evidence of hepatitis

Renal

* Creatinine < 2.0 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No ischemic cardiac disease, congestive heart failure, or myocardial infarction within the past 6 months
* No uncontrolled cardiac rhythm disturbance
* No myocardial ischemia or heart failure by exercise radionuclide scan for patients with a history of cardiac disease, significant risk factors for coronary artery disease, or ≥ 65 years of age

Pulmonary

* Pulmonary function normal by exercise radionuclide scan for patients with a history of cardiac disease, significant risk factors for coronary artery disease, or ≥ 65 years of age

Immunologic

* HIV negative
* No known hypersensitivity to the study drug, Tween-80®, or human immunoglobulin
* No uncontrolled active infection

Neurologic

* No seizure disorder
* No objective peripheral neuropathy ≥ grade 2
* No clinically significant neurologic deficit

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must consent to the placement of a central venous line OR demonstrate stable peripheral IV access
* Must be willing and able to discontinue antihypertensive medications (if advised to do so) on the days of study drug infusion
* No uncontrolled active peptic ulcer
* No known grade 4 side effects related to prior interleukin-2
* No diabetes mellitus that has required systemic therapy (e.g., oral hypoglycemic agents or insulin) within the past 3 months
* No other significant illness
* No significant psychiatric disability

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior monoclonal antibodies for biologic therapy, tumor imaging, purging of autologous bone marrow/stem cells for re-infusion, or for any other reason allowed provided there is documented absence of detectable antibody to hu14.18 by serology
* No concurrent growth factors

Chemotherapy

* No immediate requirement for palliative chemotherapy
* No concurrent anticancer chemotherapy

Endocrine therapy

* More than 2 weeks since prior and no concurrent corticosteroids (e.g., dexamethasone)
* No immediate requirement for palliative hormonal therapy

Radiotherapy

* No immediate requirement for palliative radiotherapy

  * Concurrent palliative radiotherapy to localized painful lesions allowed provided ≥ 1 measurable or evaluable lesion is not irradiated AND the irradiated lesion is not used to assess tumor response

Surgery

* More than 3 weeks since prior major surgery
* No prior organ allografts

Other

* More than 2 weeks since other prior and no concurrent immunosuppressive drugs
* No prior standard or experimental systemic therapy for stage IV melanoma
* No concurrent myelosuppressive antineoplastic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate and duration of response by clinical exam and radiology studies after every 2 courses

SECONDARY OUTCOMES:
Adverse events by clinical assessment daily during treatment and weekly after completion of study treatment
Immunologic activation induced by hu14.18-interleukin-2 after every 2 courses
Induction of anti-idiotypic antibodies on days 1, 3, 4, and 8 of each course

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Albertini, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu